CLINICAL TRIAL: NCT05858840
Title: Place of Urinary Artificial Sphincter in Children With Neurogenic Bladder
Brief Title: Urinary Artificial Sphincter in Children
Acronym: SUA
Status: Completed | Type: Observational
Sponsor: University of Lorraine (Other)
Responsible Party: Principal Investigator, Dr Christelle DESTINVAL, Principal Investigator, University of Lorraine
Other Study IDs: ULorr; 2023PI008 (Registry Identifier: DRCI)
Record Dates: First submitted 2023-04-12; First posted 2023-05-15 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Neurogenic Bladder; Bladder Dysfunction; Spina Bifida; Child, Only
Keywords: Urinary Artificial Sphincter; Neurogenic Bladder; Children; Outcomes; Retrospective Study
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Dysraphism | interventions — Urinary Sphincter, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Urinary Artificial Sphincter (UAS) in Children — Patients aged under 18 years old with UAS

SUMMARY:
Retrospective monocentric study of the outcomes of patients with neurogenic bladder, who had a urinary artificial sphincter before the age of 18 years old.

Hypothesis: what was the impact of the urinary artificial sphincter on the global management of the patient.

DETAILED DESCRIPTION:
The management of patients with neurogenic bladder is complex. Several patients have been operated multiple times. Surgical procedures such as Mitrofanoff's, bladder neck surgery, bladder augmentation and urinary artificial sphincter, are common.

The investigators want to analyse the participants data, that led to indication of an urinary artificial sphincter, and its outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were younger than 18 years old when they had an urinary artificial sphincter

Exclusion Criteria:

* Patients who were 18 years old or older when they had an urinary artificial sphincter

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients younger than 18 years old who have neurogenic bladders.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with refractory urinary incontinence | Before surgery
  Participants with urinary incontinence without response to medical treatment or catheterization
Impact of urinary artificial sphincter on the participants' incontinence | Through study completion, an average of 2 years
  Three outcomes are possible: the participant is continent, the participant is continent with catheterization or the patient is incontinent.

SECONDARY OUTCOMES:
Impact of bladder augmentation on participants' incontinence | Through study completion, an average of 2 years
  Analysing the presence of bladder augmentation in participants with urinary artificial sphincter. Three outcomes are possible: the participant is continent, the participant is continent with catheterization or the patient is incontinent.
Impact of Mitrofanoff procedure on participants' incontinence | Through study completion, an average of 2 years
  Analysing the presence of Mitrofanoff procedure in participants with urinary artificial sphincter. hree outcomes are possible: the participant is continent, the participant is continent with catheterization or the patient is incontinent.
Impact of bladder neck surgery on participants' incontinence | Through study completion, an average of 2 years
  Analysing the presence of bladder neck surgery in participants with urinary artificial sphincter. hree outcomes are possible: the participant is continent, the participant is continent with catheterization or the patient is incontinent.
Complications after urinary artificial sphincter | Through study completion, an average of 2 years
  Medical and surgical complications after urinary artificial sphincter
Operating time | Perioperatively
  Operating time
Length of stay | From the day of hospitalization to the day of discharge home, up to 20 days
  Length of stay
Last follow-up | Through study completion, an average of 2 years
  Follow-up represents the time between the surgery and postoperative consultation dates in days, months, or years. Generally, there are a-month-follow-up, a three month-follow-up, a six month-follow-up, and a year-follow-up. The surgeon can see the patient if there is any problem between these consultations. After a year of follow-up, it is up to the surgeon to decide if the patient needs to be seen yearly or not. The last follow-up date is crucial because it indicates how the patient is and if other follow-up dates need to be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Destinval, MD, Principal Investigator — University of Lorraine
Locations (1):
- ULorraine, Vandœuvre-lès-Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: No
In the name of anonymization the investigators won't share individual participant data

REFERENCES:
- [Background] Delgado-Miguel C, Munoz-Serrano A, Amesty V, Rivas S, Lobato R, Martinez-Urrutia MJ, Lopez-Pereira P. Artificial urinary sphincter in congenital neuropathic bladder: Very long-term outcomes. Int J Urol. 2022 Jul;29(7):692-697. doi: 10.1111/iju.14874. Epub 2022 Mar 26. PMID 35340070
- [Background] Sheppard KE, Roberts JL, Blum M. Adrenocorticotropin-releasing factor down-regulates glucocorticoid receptor expression in mouse corticotrope tumor cells via an adenylate cyclase-dependent mechanism. Endocrinology. 1991 Aug;129(2):663-70. doi: 10.1210/endo-129-2-663. PMID 1855464